



**Neurology Infusion and Planned Investigation Unit** 

Department of Neurology Barts and the London NHS Trust The Royal London Hospital, Ward 11D, 11th Floor, Central Tower Whitechapel, London, E1 1BB Switchboard: 020 3594 0000 www.bartsandthelondon.nhs.uk

Subject Initials:

Subject Identification Number:

## PATIENT CONSENT FORM FOR PRESENT USAGE AND FOR STORAGE AND FUTURE USE OF SAMPLES

## Oral Cladribine B-cell study (Clad-B study) (IRAS project ID: 262436)

| | Please initial box: | | | Yes | No |
|---|---|---|---|---|---|
| 1. | I confirm that I have read and understand the Patient Information Sheet dated 28 <sup>th</sup> May 2019 for the above study and have had the opportunity to ask questions. Questions have been answered to my satisfaction. | | | | |
| 2. | I agree that my cerebrospinal spinal this study. | rospinal spinal fluid (CSF), urine and blood samples may be used for | | | |
| 3. | I agree that these samples will be stored in the Blizard Institute, Queen Mary University London, and may be used in future ethically approved projects, as described in the information sheet. | | | | |
| 4. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. If I withdraw from this study then I understand it is my right to ask for any stored samples to be destroyed. The data collected up to the point of withdrawal will be included in the analysis at the end. | | | | |
| 5. | I understand that sections of my medical notes and data collected during the study may be looked at by authorised persons in the research team where it is relevant to my taking part in this research. Barts Health NHS Trust is the sponsor for this study based in the United Kingdom. We will be using information from you and your medical records in order to undertake this study and will act as the data controller for this study. Barts Health NHS Trust and regulatory organisations may look at your medical and research records to check the accuracy of the research study. I give permission for these individuals to have access to my records. | | | | |
| 6. | I agree to take part in the above study. | | | | |
| 7. | I agree my GP will be informed of my participation in this study | | | | |
| <br>Nam | e of Patient | Signature | Date | | |
| <br>Rese | archer | Signature | Date | | |